CLINICAL TRIAL: NCT06588855
Title: A Phase III, Multicenter, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Induction Therapy With RO7790121 in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Assess the Efficacy and Safety of Induction Therapy With Afimkibart (Also Known as RO7790121) in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: Ametrine-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA45330; 2024-513015-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Moderately to Severely Active Ulcerative Colitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afimkibart (Experimental): Participants will receive afimkibart intravenously (IV) followed by afimkibart subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Placebo (Placebo Comparator): Participants will receive placebo IV followed by placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afimkibart — Participants will receive afimkibart IV followed by afimkibart subcutaneous SC injection.
  Other Names: PF-06480605; RVT-3101; RG6631; RO7790121
  Arms: Afimkibart
Drug: Placebo — Placebo matching IV afimkibart. Placebo matching SC afimkibart.
  Arms: Placebo

SUMMARY:
This Phase III, multicenter, double-blind, placebo-controlled study will evaluate the efficacy and safety of induction therapy with Afimkibart (RO7790121) compared with placebo in participants with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UC
* Moderately to severely active UC assessed by mMS
* Bodyweight >= 40 kilogram (kg)
* Up to date with colorectal cancer (CRC) screening performed according to local standards
* Demonstrated inadequate response, loss of response and/or intolerance to at least one protocol-specified conventional or advanced UC therapy
* Males and females of childbearing potential must meet protocol criteria for contraception requirements

Exclusion Criteria:

* Currently known complications of UC (e.g. fulminant colitis, toxic megacolon)
* Current diagnosis of Crohn's disease (CD) or indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis
* Presence of an ostomy or ileoanal pouch
* Current diagnosis or suspicion of primary sclerosing cholangitis
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Past or current evidence of definite low-grade or high-grade colonic dysplasia or adenomas or neoplasia not completely removed
* History of malignancy within 5 years, with the exception of malignancies adequately treated with resection for non-metastatic basal cell or squamous cell cancer or in situ cervical cancer
* Evidence of infection with Clostridioides difficile (C. difficile; formerly known as Clostridium difficile), cytomegalovirus (CMV), human immunodeficiency virus (HIV), Hepatitis B (HBV), Hepatitis C (HCV)
* Has evidence of active tuberculosis (TB), latent TB not successfully treated (per local guidance) or inadequately treated TB
* Has received protocol-specified prohibited medicines, including known exposure to any type of anti-TL1A therapy

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission | At Week 12
  Percentage of participants achieving Modified Mayo Score (mMS) <=2 with stool frequency subscore (SFS) = 0 or 1 (up to 1-2 stools more than normal), rectal bleeding subscore (RBS) = 0 (no blood seen) and endoscopic subscore (ES) = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.

SECONDARY OUTCOMES:
Change in Partial Modified Mayo Score (pmMS) | From baseline to Week 2
  Change in pmMS from baseline to Week 2. pmMS is a composite score of ulcerative colitis signs and symptoms activity given by the sum of the SFS and RBS. SFS is measured on a scale from 0 (normal number of stools) to 3 (5 or more stools than normal). RBS is measured on a scale from 0 (no blood seen) to 3 (blood alone passed).
Percentage of Participants with Endoscopic Improvement | At Week 12
  Percentage of participants achieving endoscopic subscore of 0 or 1 (normal appearance of mucosa or mild disease) at Week 12.
Percentage of Participants with Endoscopic Remission | At Week 12
  Percentage of participants achieving endoscopic subscore of 0 (normal appearance of mucosa) at Week 12.
Percentage of Participants with Clinical Response | At Week 12
  Percentage of participants achieving a decrease in mMS of at least 2 points and 30% from baseline and either a decrease in RBS >= 1 or RBS = 0 or 1 (no blood seen or stool with streaks of blood) at Week 12. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. SFS is measured on a scale from 0 (normal number of stools) to 3 (5 or more stools than normal). RBS is measured on a scale from 0 (no blood seen) to 3 (blood alone passed). ES is measured on a scale from 0 (normal appearance of mucosa) to 3 (severe disease).
Percentage of Participants with Histologic Improvement | At Week 12
  Percentage of participants achieving a histologic improvement, defined as Geboes <=3.1 at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Histologic Remission | At Week 12
  Percentage of participants achieving a histologic remission, defined as Geboes <2B at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Participants with Histologic-Endoscopic Mucosal Improvement | At Week 12
  Percentage of participants achieving Geboes <= 3.1 and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Histologic-Endoscopic Remission | At Week 12
  Percentage of participants achieving Geboes < 2 and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Clinical Remission: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving mMS <= 2 with SFS = 0 or 1 (up to 1-2 stools more than normal), RBS = 0 (no blood seen) and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12 in biomarker-defined subgroups. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.
Percentage of Participants with Endoscopic Improvement: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving endoscopic subscore of 0 or 1 (normal appearance of mucosa or mild disease) at Week 12 in biomarker-defined subgroups.
Change in Bowel Urgency | Baseline through Week 12
  Change in bowel urgency from baseline through Week 12. Bowel urgency is measured on a scale from 0 (None) to 4 (Severe).
Change in Abdominal Pain | Baseline through Week 12
  Change in abdominal pain from baseline through Week 12. Abdominal pain is measured on a scale from 0 (None) to 4 (Severe).
Change in Fatigue | Baseline to Week 12
  Change in fatigue as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) from baseline to Week 12. FACIT-Fatigue is a 13-item self-reported assessment of the level and impact of fatigue. The overall FACIT-Fatigue score ranges between 0 and 52, with higher scores associated with better quality of life concerns related to fatigue.
Change in Health-Related Quality of Life | Baseline to Week 12
  Change in Inflammatory Bowel Disease Questionnaire (IBDQ) score from baseline to Week 12. IBDQ is a 32-item self-reported assessment of health-related quality of life in participants with inflammatory bowel disease. The overall IBDQ score ranges from 32 to 224, with higher scores associated with better health-related quality of life.
Overall Change in UC Symptoms | Baseline to Week 2 and Week 12
  Patient Global Impression of Change (PGIC) from baseline to Weeks 2 and 12. PGIC measures overall change in ulcerative colitis symptoms from "Much better" to"Much worse".
Overall Severity in UC Symptoms | Baseline to Week 2 and Week 12
  Patient Global Impression of Severity (PGIS) from baseline to Weeks 2 and 12. PGIS measures severity of ulcerative colitis symptoms from "None" to "Very severe".
Incidence and Severity of Adverse Events (AEs) | Up to 30 Weeks after Baseline
  Incidence and severity of AEs, including serious AEs, AEs leading to treatment discontinuation and AEs of special interest.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (189):
- United States (62):
  - Mayo Clinic Hospital, Scottsdale, Arizona
  - Arizona Digestive Health, P.C (ADH), Sun City, Arizona
  - Om Research LLC, Apple Valley, California
  - Valley View Internal Medicine, Garden Grove, California
  - Gastro Care Associates, Lancaster, California
  - Hoag Memorial Hospital Presbyterian;Hoag Center for Research and Education, Newport Beach, California
  - Hi Tech and Global Research, LLC, Coral Gables, Florida
  - The Sister Life Research, Hialeah, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Ambert Medical Research, Miami, Florida
  - Gastroenterology Institute of Orlando, Orlando, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - University of South Florida School of Medicine Morsani Center for Advanced Health Care, Tampa, Florida
  - Guardian Angel Research Center, LLC, Tampa, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Randomize Now, LLC, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Illinois Gastroenterology Group-Glenview powered by GI Alliance, Glenview, Illinois
  - GI Alliance - Gurnee, Gurnee, Illinois
  - Gastro Health Partners, LLC, New Albany, Indiana
  - Kansas Gastroenterology, LLC under Clinical Trials Network, Wichita, Kansas
  - One GI: GHP - Gastroenterology Health Partners Louisville, Louisville, Kentucky
  - Louisiana Research Center - GastroIntestinal Associates, Shreveport, Louisiana
  - Delta Gastroenterology & Endoscopy Center, Southaven, Mississippi
  - Ellipsis Research Group, Brooklyn, New York
  - Weill Cornell Medical College, New York, New York
  - DiGiovanna Inst for Med Ed&Res, North Massapequa, New York
  - Queens Village Medical Care, Queens Village, New York
  - Gastroenterology Group Of Rochester, LLP, Rochester, New York
  - James J Peters Veterans Administration Medical Center - NAVREF, The Bronx, New York
  - Charlotte Gastroenterology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Omega Research North Carolina, LLC, Fuquay-Varina, North Carolina
  - Peters Medical Research (PMR), LLC, High Point, North Carolina
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - University of Cincinnati Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Gastroenterology Group, Columbus, Ohio
  - Ohio State University, Hilliard, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, Westlake, Ohio
  - Frontier Clinical Re search, LLC, Uniontown, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastroenterology Associates, Greenville, South Carolina
  - Gastro One, Cordova, Tennessee
  - Uni of Texas Medical Branch, Galveston, Texas
  - GI Alliance, Garland, Texas
  - Amel Med LLC, Georgetown, Texas
  - Cano Medical Center, Harlingen, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - Integrity Advanced Therapeutics PLLC, Houston, Texas
  - GI Alliance - Bay Area Gastroenterology, Lubbock, Texas
  - TDDC dba GI Alliance Research, Mansfield, Texas
  - Southern Star Research Institute, LLC., San Antonio, Texas
  - Baylor Scott and White Medical Center, Temple, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Gastroenterology Consultants of SWVA, Roanoke, Virginia
- Argentina (2):
  - Hospital Britanico, Ciudad Autonoma Bs As
  - Instituto Medico CER, Quilmes
- Australia (4):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Coral Sea Clinical Research Institute, Mackay, Queensland
  - Footscray Hospital, Footscray, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (4):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - CHU St Pierre (St Pierre), Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - AZ Oostende, Ostend
- Brazil (6):
  - Instituto Lobus Unimed Volta Redonda, Volta Redonda, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Newdata Clinical Trials, Aracaju, Sergipe
  - CECIP - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Centro Paulista de Investigacao Clinica - CEPIC, São Paulo, São Paulo
- Bulgaria (3):
  - Second Multiprofile Hospital For Active Treatment-Sofia, Sofia Town, Sofia
  - MC " Sveti Ivan Rilski Chudotvorets- 2010, Plovdiv
  - "City Clinic UMHAC" EOOD, Sofia
- Canada (5):
  - Barrie GI Associates, Barrie, Ontario
  - GNRR Digestive Clinics and Research Center Inc., Brampton, Ontario
  - London Health Sciences Centre Uni Campus, London, Ontario
  - TIDHI Innovation Inc., Toronto, Ontario
  - CIUSSS-de-l?Est-de-l?Île-de-Montréal, Montreal, Quebec
- Centro de Investigación Clínica UC-CICUC, Santiago, Chile
- China (18):
  - Beijing No.6 Hospital, Beijing, Beijing Municipality
  - The First Affilliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Third Xiangya Hospital Centrel South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Guangzhou First People's Hospital, Guangzhou
  - The second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Huizhou Central People's Hospital, Huizhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - First Affiliated Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhongshan Hospital Xiamen University, Xiamen
- Croatia (2):
  - Borzan Polyclinic, Osijek
  - Clinical Hospital Center Sestre Milosrdnice, Zagreb
- Czechia (3):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - ISCARE a.s., Prague
- Ålborg Universitets Hospital, Aalborg, Denmark
- France (5):
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - CHU Clermont Ferrand - Hôtel Dieu, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Polyclinique Grand Sud, Nîmes
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg
  - Medizinisches Zentrum Klinikum Lueneburg, Lüneburg
  - Klinikum Ernst von Bergmann, Potsdam
- Hungary (5):
  - Észak-Pesti Centrumkórház-Honvédkórház, Budapest
  - Semmelweis Egyetem, Budapest
  - Vasutegeszsegugyi Kft. - Debreceni Egeszsegugyi Kozpont, Debrecen
  - Fejer Varmegyei Szent György Egyetemi Oktatokorhaz, Székesfehérvár
  - Vas-Oxy Egeszsegugyi Kft, Szombathely
- India (8):
  - Surat Institute of Digestive Sciences Hospitals, Surat, Gujarat
  - Gujarat Gastro and Vascular Hospital, Surat, Gujarat
  - MIDAS Multispeciality Hospital, Nagpur (urban), Maharashtra
  - Sahyadri Super Speciality Hospital, Nashik, Maharashtra
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - SMS Superspeciality Hospital, Jaipur, Rajasthan
  - AIG Hospitals, Gachibowli, Telangana
  - Yashoda Hospitals, Secunderabad, Telangana
- Israel (2):
  - Soroka Medical Center, Beersheba
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (8):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi-Via Massarenti, Bologna, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico Di Roma, Rome, Lazio
  - Ospedale Isola Tiberina Gemelli, Rome, Lazio
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Azienda Ospedaliera San Gerardo di Monza, Monza MI, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
- Mexico (2):
  - Boca Clinical Trials Mexico S.C. (Cd. Mexico), Miguel Hidalgo, Mexico CITY (federal District)
  - FAICIC S de R.L. de C.V, Veracruz
- ETZ Elisabeth, Tilburg, Netherlands
- Poland (19):
  - Szpital Zakonu Bonifratrow Sw. Jana Bozego w Lodzi sp. z o.o., ?ód?
  - Gastromed Kralisz, Romatowski, Stachurska sp.j., Bia?ystok
  - Medical Center Kermed, Bydgoszcz
  - Szpital Miejski sw. Jana Paw?a II w Elblagu, Elblag
  - Centrum Medyczne CLW-med Aneta Cichomska , Joanna Luka -Wendrowska, Grudzadz
  - Osrodek Badan Klinicznych Bd Research, I?awa
  - MZ Badania Slowik Zymla Sp.j., Knurów
  - Centrum Medyczne Promed, Krakow
  - Medrise sp z o.o, Lublin
  - Clinical Research Center Sp. z o.o. MEDIC-R Spó?ka Komandytowa, Poznan
  - EMC Instytut Medyczny SA, Późna
  - Gabinety Lekarskie Rivermed, Późna
  - Endoskopia Sp. z o.o., Sopot
  - Sonomed Sp. z o.o., Szczecin
  - Centrum Zdrowia-MDM, Warsaw
  - Medon Clinical Research sp. z o.o, Warsaw
  - Vivamed Spolka Z Ograniczona Odpowiedzialnoscia, Warsaw
  - PlanetMed sp. z o.o., Wroc?aw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (6):
  - Hospital de Braga, Braga
  - Hospital da Luz Lisboa, Lisbon
  - Centro Hospitalar do Algarve - Hospital de Portimao, Portimão
  - Hospital de Sao Joao, Porto
  - Centro Hospitalar de Entre Douro e Vouga - H. São Sebastião, Santa Maria da Feira
  - Hospital Sao Teotonio, Viseu
- Klinical Investigations Group LLC, San Juan, Puerto Rico
- General Hospital "Djordje Joanovic", Zrenjanin, Serbia
- Slovakia (2):
  - KM Management spol. s r.o., Nitra
  - Accout Center s.r.o., Šahy
- Spain (3):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinico Univ. Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- China Medical University Hospital, Taichung, Taiwan
- Thailand (3):
  - Division of Gastroenterology, Depart of Internal Med., Fac of Med., Chiang Mai University, Chiang Mai
  - Burapha University Hospital, Chon Buri
  - Sunpasitthiprasong Hospital, Ubonratchathani
- United Kingdom (6):
  - Leicester General Hospital, Leicester
  - Bronglais General Hospital, Llanrhystud
  - King College Hospital NHS Foundation Trust, London
  - Peterborough City Hospital, Peterborough
  - Stepping Hill Hospital, Stockport
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing